CLINICAL TRIAL: NCT00270101
Title: A Placebo-Controlled Study on the Effect of r-huEPO in Patients With Multiple Myeloma Followed by an Open-Label Extension
Brief Title: The Effect of Epoetin Alfa on the Anemia of Patients With Multiple Myeloma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR005911
Record Dates: First submitted 2005-12-22; First posted 2005-12-26 (Estimated); Last update posted 2011-05-18 (Estimated); Status verified 2011-01

CONDITIONS: Anemia; Multiple Myeloma
Keywords: anemia; cancer; quality of life; chemotherapy; hemoglobin; multiple myeloma; transfusion; epoetin alfa; epoetin; erythropoietin
MeSH Terms: conditions — Anemia; Multiple Myeloma; Neoplasms | interventions — Epoetin Alfa

INTERVENTIONS:
Drug: epoetin alfa

SUMMARY:
The purpose of this study is to evaluate the safety and effectiveness of epoetin alfa versus placebo in reducing the transfusion requirements in anemic patients with multiple myeloma, and to investigate the quality-of-life benefits associated with the use of epoetin alfa. Epoetin alfa is a genetically engineered protein that stimulates red blood cell production.

DETAILED DESCRIPTION:
Cancer patients often experience anemia due to the disease itself, chemotherapy or both. Quality of life is also affected, in part because of the fatigue associated with anemia. Previous studies with epoetin alfa have suggested that achieving a higher hemoglobin level may improve quality of life and help patients live longer. This study is a 12-week randomized, double-blind, placebo-controlled, multicenter study (with an open-label extension) to assess the effectiveness of treatment with epoetin alfa in reducing the need for red cell transfusion by improving anemia in patients with multiple myeloma whose hemoglobin is less than 11 grams per deciliter. There will be 4 groups of patients in the study. Patients will first be placed into 2 groups according to whether or not they received at least 1 blood transfusion within the previous 3 months. Within each of these 2 groups, patients will then be randomly assigned to receive either epoetin alfa or placebo for 12 weeks. Dosing is initiated at 150 units per kilogram (U/kg) injected under the skin 3 times weekly for 4 weeks, then either continued at 150 U/kg or adjusted to 300 U/kg according to hemoglobin levels for the remaining 8 weeks. All patients who complete the 12-week double-blind period will be eligible to continue receiving epoetin alfa for an additional 12 weeks in an open-label extension of the study. The primary measures of effectiveness will be determined by the number of units of blood transfused, the proportion of patients requiring transfusion, and the number of units transfused relative to whether or not they received transfusions before the study. Additional effectiveness measures include the number of patients whose hemoglobin level reach at least 12 grams per deciliter (anemia considered "corrected") or who have an increase in hemoglobin of at least 2 grams per deciliter, and the change in the percentage of red blood cells and number of developing red blood cells in the blood. Changes in quality-of-life (Nottingham and visual analog scale) and performance scores will also be measured. Safety evaluations (incidence of adverse events, laboratory tests, and vital signs) and changes in underlying multiple myeloma will be assessed. The hypothesis of the study is that epoetin alfa will be superior to placebo in reducing the need for transfusions and improving anemia and quality of life. Double-blind: Epoetin alfa 150 units per kilogram (U/kg) injected under the skin 3 times weekly for 4 weeks; then either continued at 150 U/kg or adjusted to 300 U/kg according to hemoglobin levels for the remaining 8 weeks. Open-label: dose to maintain target hemoglobin range.

ELIGIBILITY:
Inclusion Criteria:

* Patients with documented multiple myeloma defined by standard criteria, with at least 6 months having elapsed since beginning chemotherapy
* having a self-care performance score of 0, 1, 2, or 3 (patients' ability to perform daily activities, a score ranging from 0 [fully active, no disease restriction] to 3 [capable of only limited self-care, confined to bed or chair more than 50% of waking hours])
* having a life expectancy of at least 3 months
* having a baseline hemoglobin <11 g/dL and baseline count of <100,000 microliter for developing red cells
* with an ability to administer self-injections

Exclusion Criteria:

* Patients having clinically significant disease other than cancer
* having evidence of uncontrolled hypertension or a history of seizure
* having untreated iron, folate, or Vitamin B12 deficiency
* receiving a transfusion within 7 days of study entry, or androgen therapy within 1 month of study entry
* receiving dialysis at baseline screening

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Actual)
Dates: Start 1995-01; Study Completion 1996-09 (Actual)

PRIMARY OUTCOMES:
Proportion of patients requiring transfusion and number of units transfused relative to whether or not patients received transfusion(s) before the study.

SECONDARY OUTCOMES:
Increase in hemoglobin, hematocrit, developing red blood cells in the blood; Changes in quality-of-life; Safety evaluations (incidence of adverse events, laboratory tests, and vital signs) including changes in underlying multiple myeloma.

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.

REFERENCES:
- See also: The effect of epoetin alfa on the anemia of patients with multiple myeloma — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=682&filename=CR005911_CSR.pdf